CLINICAL TRIAL: NCT06126952
Title: Randomized, Double-blind, Cross-over Clinical Trial to Assess Onset of Action and Efficacy of Azelastine Hydrochloride 0.15% Nasal Spray in the Treatment of Allergen-Induced Allergic Rhinitis Symptoms in an Environmental Exposure Unit in Comparison to Placebo and Mometasone Furoate/Olopatadine Hydrochloride Nasal Spray
Brief Title: Azelastine Allergen Chamber - Onset of Action Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AZEL-NS-2001; C2D03217 (Other: Cliantha Research, Canada)
Record Dates: First submitted 2023-10-27; First posted 2023-11-13 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Nasal Sprays; azelastine; Mometasone Furoate

STUDY DESIGN:
Intervention Model Description: The study will be a single-center, randomized, placebo-controlled, double-blind trial with three periods and six sequences (cross-over design).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Treatment A (Azelair)+Treatment B (Placebo)+Treatment C (Ryaltris), min. 14 days wash-out period (Experimental): Cross-over design
  Interventions: Drug: Treatment A: Azelastine hydrochloride 0.15% nasal spray (Azelair); Drug: Treatment B: Placebo (Azelastine 0.15% vehicle) nasal spray; Drug: Treatment C: Ryaltris (Active Control) - mometasone furoate monohydrate and olopatadine hydrochloride nasal spray
- Treatment B (Placebo)+Treatment C (Ryaltris)+Treatment A (Azelair), min. 14 days of wash-out period (Experimental): Cross-over design
  Interventions: Drug: Treatment A: Azelastine hydrochloride 0.15% nasal spray (Azelair); Drug: Treatment B: Placebo (Azelastine 0.15% vehicle) nasal spray; Drug: Treatment C: Ryaltris (Active Control) - mometasone furoate monohydrate and olopatadine hydrochloride nasal spray
- Treatment C (Ryaltris)+Treatment A (Azelair)+Treatment B (Placebo), min. 14 days of wash-out period (Experimental): Cross-over design
  Interventions: Drug: Treatment A: Azelastine hydrochloride 0.15% nasal spray (Azelair); Drug: Treatment B: Placebo (Azelastine 0.15% vehicle) nasal spray; Drug: Treatment C: Ryaltris (Active Control) - mometasone furoate monohydrate and olopatadine hydrochloride nasal spray
- Treatment A (Azelair)+Treatment C (Ryaltris)+Treatment B (Placebo), min. 14 days of wash-out period (Experimental): Cross-over design
  Interventions: Drug: Treatment A: Azelastine hydrochloride 0.15% nasal spray (Azelair); Drug: Treatment B: Placebo (Azelastine 0.15% vehicle) nasal spray; Drug: Treatment C: Ryaltris (Active Control) - mometasone furoate monohydrate and olopatadine hydrochloride nasal spray
- Treatment B (Placebo)+Treatment A (Azelair)+Treatment C (Ryaltris), min.14 days of wash-out period (Experimental): Cross-over design
  Interventions: Drug: Treatment A: Azelastine hydrochloride 0.15% nasal spray (Azelair); Drug: Treatment B: Placebo (Azelastine 0.15% vehicle) nasal spray; Drug: Treatment C: Ryaltris (Active Control) - mometasone furoate monohydrate and olopatadine hydrochloride nasal spray
- Treatment C (Ryaltris)+Treatment B (Placebo)+Treatment A (Azelair), min. 14 days of wash-out period (Experimental): Cross-over design
  Interventions: Drug: Treatment A: Azelastine hydrochloride 0.15% nasal spray (Azelair); Drug: Treatment B: Placebo (Azelastine 0.15% vehicle) nasal spray; Drug: Treatment C: Ryaltris (Active Control) - mometasone furoate monohydrate and olopatadine hydrochloride nasal spray

INTERVENTIONS:
Drug: Treatment A: Azelastine hydrochloride 0.15% nasal spray (Azelair) — 2 sprays per nostril of Azelastine 0.15% twice daily.
  Total dose of active drug:
  1644 mcg azelastine hydrochloride per day
Drug: Treatment B: Placebo (Azelastine 0.15% vehicle) nasal spray — 2 sprays per nostril of Placebo twice daily.
Drug: Treatment C: Ryaltris (Active Control) - mometasone furoate monohydrate and olopatadine hydrochloride nasal spray — 2 sprays per nostril of Ryaltris twice daily.
  Total dose of active drug:
  200 mcg mometasone furoate and 4800 mcg olopatadine per day

SUMMARY:
This study is to assess the Onset of Action and Efficacy of azelastine hydrochloride 0.15% in treating the nasal symptoms of seasonal allergic rhinitis (SAR) induced by an allergen challenge in an Environmental Exposure Unit (EEU) followed by a single dose and a 3-day treatment at home.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female subjects (childbearing and non-childbearing potential, non-childbearing potential defined as females with no menstruation for at least 1 year at screening and documented FSH > 35 IU/L) aged 18 to 55 years (inclusive) at screening.
* History of SAR to ragweed pollen for at least the previous 2 ragweed pollen seasons.
* Positive skin prick test (SPT) response to ragweed pollen (allergen induced wheal diameter at least 3 mm larger than the negative control). A test performed at Cliantha Research in the previous 12 months may be used to qualify the subject.

Main Exclusion Criteria:

Safety Concerns:

* History of allergic reaction to azelastine hydrochloride, olopatadine hydrochloride, mometasone furoate, or one of the excipients / components of the study treatments
* History of anaphylaxis, cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, metabolic, psychiatric, neurological, or other disease at screening that may affect subject safety during the study or evaluation of the study endpoints at the discretion of the Investigator and/or designee.
* Subjects with a current diagnosis of asthma or subjects with measured forced expiratory volume in 1 second (FEV1) <75% of the predicted value using Global Lung Function Initiative set from 2012 for references.
* Pregnant, breast-feeding, or planning a pregnancy during the study and women of childbearing potential not using adequate contraception.

Lack of suitability for the study:

* Use of prohibited therapies as specified in the respective table of the protocol.
* Acute or chronic sinusitis or non-allergic rhinitis, at the discretion of the Investigator and/or designee.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in TNSS at each post-dose assessment time point (0 to 4 hours after a single dose). | 0 to 4 hours post application
  Onset of action of azelastine hydrochloride 0.15% nasal spray (Azelastine 0.15%) in treating the nasal symptoms of seasonal allergic rhinitis (SAR) induced by an allergen challenge in an Environmental Exposure Unit (EEU), measured by a difference from placebo in the change from baseline in patient -assessed instantaneous Total nasal symptom score (TNSS).
  FDA guideline defines onset of action as the first time point after initiation of treatment when the product demonstrated a greater change from baseline compared to placebo which proved durable.
  The TNSS is comprised of 4 symptoms from the nose, each scored on a scale of 0 to 3 (0 = none and 3 = severe). The sum of the TNSS contributes to a score ranging from 0 - 12.

SECONDARY OUTCOMES:
Changes from baseline in TNSS at each post-dose assessment time point (0 to 4 hours after a single dose) at Visits 3, 6, and 9. | 0 to 4 hours post application
  Onset of action, measured by the differences of both active treatments versus placebo in the change from baseline in patient-assessed instantaneous total symptom scores following treatment.
  FDA guideline defines onset of action as the first time point after initiation of treatment when the product demonstrated a greater change from baseline compared to placebo which proved durable.
  The TNSS is comprised of 4 symptoms from the nose, each scored on a scale of 0 to 3 (0 = none and 3 = severe). The sum of the TNSS contributes to a score ranging from 0 - 12.
Changes from baseline in TOSS at each post-dose assessment time point (0 to 4 hours after a single dose) at Visits 3, 6, and 9. | 0 to 4 hours post application
  Onset of action, measured by the differences of both active treatments versus placebo in the change from baseline in patient-assessed instantaneous total symptom scores following treatment.
  FDA guideline defines onset of action as the first time point after initiation of treatment when the product demonstrated a greater change from baseline compared to placebo which proved durable.
  The TOSS is comprised of 3 symptoms from the eyes, each scored on a scale of 0 to 3 (0 = none and 3 = severe). The sum of the TOSS contributes to a score ranging from 0 - 9.
Changes from baseline in T7SS at each post-dose assessment time point (0 to 4 hours after a single dose) at Visits 3, 6, and 9. | 0 to 4 hours post application
  Onset of action, measured by the differences of both active treatments versus placebo in the change from baseline in patient-assessed instantaneous total symptom scores following treatment.
  FDA guideline defines onset of action as the first time point after initiation of treatment when the product demonstrated a greater change from baseline compared to placebo which proved durable.
  The total 7 symptoms score (T7SS) will be the combination of the TNSS and TOSS, for a combined maximum score of 21.
Change from baseline in individual symptom scores at each post-dose assessment time point (0 to 4 hours after a single dose) at Visits 3, 6, and 9. | 0 to 4 hours post application
  Onset of action, measured by change from baseline in individual symptom scores at each post-dose assessment time point (0 to 4 hours after a single dose) at Visits 3, 6, and 9.
  Each individual symptom is scored on a scale of 0 to 3 (0 = none and 3 = severe).
  Secondary endpoint include pairwise treatment comparisons of both active treatments versus placebo.
Changes from baseline in TNSS for all assessment time-points together. | 0 to 4 hours post application
  Overall Efficacy, measured by changes from baseline in TNSS for all assessments during 0-4 hours and for visits 3, 6 and 9 together.
  The TNSS is comprised of 4 symptoms from the nose, each scored on a scale of 0 to 3 (0 = none and 3 = severe). The sum of the TNSS contributes to a score ranging from 0 - 12.
Changes from baseline in TOSS for all assessment time-points together. | 0 to 4 hours post application
  Overall Efficacy, measured by changes from baseline in TOSS for all assessments during 0-4 hours and for visits 3, 6 and 9 together.
  The TOSS is comprised of 3 symptoms from the eyes, each scored on a scale of 0 to 3 (0 = none and 3 = severe). The sum of the TOSS contributes to a score ranging from 0 - 9.
Changes from baseline in T7SS for all assessment time-points together. | 0 to 4 hours post application
  Overall Efficacy, measured by changes from baseline in T7SS for all assessments during 0-4 hours and for visits 3, 6 and 9 together.
  The total 7 symptoms score (T7SS) will be the combination of the TNSS and TOSS, for a combined maximum score of 21.
Change from baseline in individual symptom scores for all assessment time-points together. | 0 to 4 hours post application
  Overall Efficacy, measured by change from baseline in individual symptom scores for all assessments during 0-4 hours and for visits 3, 6 and 9 together.
  Each individual symptom is scored on a scale of 0 to 3 (0 = none and 3 = severe).
Changes from baseline in TNSS for all assessment time-points together. | 0-4 hours after 3-day treatment
  Overall Efficacy, measured by changes from baseline in TNSS for all assessments during 0-4 hours and for visits 4, 7 and 10 together after 3-day treatment.
  The TNSS is comprised of 4 symptoms from the nose, each scored on a scale of 0 to 3 (0 = none and 3 = severe). The sum of the TNSS contributes to a score ranging from 0 - 12.
Changes from baseline in TOSS for all assessment time-points together. | 0-4 hours after 3-day treatment
  Overall Efficacy, measured by changes from baseline in TOSS for all assessments during 0-4 hours and for visits 4, 7 and 10 together after 3-day treatment.
  The TOSS is comprised of 3 symptoms from the eyes, each scored on a scale of 0 to 3 (0 = none and 3 = severe). The sum of the TOSS contributes to a score ranging from 0 - 9.
Changes from baseline in T7SS for all assessment time-points together. | 0-4 hours after 3-day treatment
  Overall Efficacy, measured by changes from baseline in T7SS for all assessments during 0-4 hours and for visits 4, 7 and 10 together after 3-day treatment.
  The total 7 symptoms score (T7SS) will be the combination of the TNSS and TOSS, for a combined maximum score of 21.
Change from baseline in individual symptom scores for all assessment time-points together. | 0-4 hours after 3-day treatment
  Overall Efficacy, measured by change from baseline in individual symptom scores for all assessments during 0-4 hours and for visits 4, 7 and 10 together after 3-day treatment.
  Each individual symptom is scored on a scale of 0 to 3 (0 = none and 3 = severe).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Couroux, Dr., Principal Investigator — Cliantha Research
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No